CLINICAL TRIAL: NCT05924841
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-B01D1 Monotherapy, SI-B003 Monotherapy and BL-B01D1+SI-B003 Combination Therapy (BL-B01D1+SI-B003) in Patients With Extensive Stage Small Cell Lung Cancer (SCLC)
Brief Title: A Study of BL-B01D1, SI-B003 and BL-B01D1+SI-B003 in Patients With Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-02
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received BL-B01D1 monotherapy, SI-B003 monotherapy or BL-B01D1 plus SI-B003 dual therapy in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — Administration by intravenous infusion

SUMMARY:
This phase II study is designed to investigate the efficacy and safety of BL-B01D1 monotherapy, SI-B003 monotherapy, and BL-B01D1+SI-B003 combination therapy in patients with extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects voluntarily participated in the study and signed informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG 0-1;
5. Patients with extensive-stage small-cell Lung cancer confirmed by histopathology and/or cytology (according to Veterans Administration Lung Study Group (VALG) staging);

   1. Cohort_A cohort of patients with extensive-stage small cell lung cancer who had failed or were intolerant to 3 or more lines of systemic antitumor therapy. The so-called intolerance refers to the patients who have received standard treatment and have grade 3-4 adverse reactions, and the patients refuse to continue the original regimen.
   2. Cohort_B Stage I subjects with previous failure or intolerance to standard therapy for extensive-stage small cell lung cancer;
   3. Cohort_B Stage II patients who have not received any previous systemic anti-tumor therapy for extensive-stage small cell lung cancer;
6. Consent to provide archival tumor tissue specimens (10 unstained sections (anti-slip) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If participants cannot provide tumor tissue samples, they can be enrolled if they meet other inclusion and exclusion criteria, after the evaluation of the investigator;
7. Must have at least one measurable lesion according to RECIST v1.1 definition; Lesions that had been previously treated with radiation could be included in a measurable lesion only if there was definite disease progression after radiation therapy.
8. Organ function level must meet the following criteria:

   1. Blood routine: hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (NEUT) ≥ 1.5×10 9 /L; Platelet count (PLT) ≥ 100×10 9 /L;
   2. Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula).
   3. Liver function: total bilirubin (TBIL≤1.5 ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were all ≤2.5 ULN, and AST and ALT were both ≤5.0 ULN when liver metastasis was present;
   4. coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5ULN;
   5. no severe cardiac dysfunction with left ventricular ejection fraction ≥50%;
   6. proteinuria ≤2+ or ≤1000mg/24h;
9. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic laboratory abnormalities such as ALP elevation, hyperuricemia, and hyperglycemia, as judged by the investigator, and toxicity without safety risk, such as alopecia, grade 2 peripheral neurotoxicity, or decreased hemoglobin ≥90g/L, as judged by the investigator);
10. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the whole treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Previous treatment with EGFR and HER3 monoclonal antibodies;
2. Antineoplastic therapy, including chemotherapy, biologic therapy, immunotherapy, definitive radiotherapy, major surgery (investigator-defined), or targeted therapy (including small-molecule tyrosine kinase inhibitors), has been administered within 4 weeks or 5 half-life cycles (whichever is shorter) before the first dose; Oral fluorouracil drugs such as S-1, capecitabine, or palliative radiotherapy within 2 weeks before the first dose;
3. Cohort_B Stage II patients who had received any previous systemic therapy for extensive-stage SCLC were not eligible for the study;
4. Cohort_B with a history of immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis, excluded;
5. Cohort_B with history of use of immunomodulatory drugs (including but not limited to thymosin, interleukin-2, interferon, etc.) within 14 days before the first dose of study drug was excluded.
6. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias or Ⅲ degree atrioventricular block requiring clinical intervention;
   2. prolonged QT interval at rest (QTc > 450 msec in men or QTc > 470 msec in women);
   3. myocardial infarction, unstable angina, cardiac angioplasty or stent implantation, coronary artery/peripheral artery bypass grafting, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident, or transient ischemic attack within 6 months before the first dose;
7. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory intestinal diseases and Hashimoto's thyroiditis, etc., excluding type I diabetes mellitus, hypothyroidism that can be controlled only by replacement therapy, and skin diseases without systemic treatment (such as vitiligo and psoriasis);
8. Other malignant tumors that have progressed or require treatment within 5 years before the first dose, except for radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, radical resection of carcinoma in situ, such as carcinoma in situ of the breast, and prostate cancer; Notes: Patients with localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and PSA < 10ng/mL at prostate cancer diagnosis (as measured) who had received radical treatment and no biochemical recurrence of prostate specific antigen (PSA) were eligible to participate in this study).
9. A history of (non-infectious) interstitial lung disease (ILD)/pulmonary inflammation requiring steroid treatment, or current ILD/ pulmonary inflammation, or suspected ILD/ pulmonary inflammation that cannot be ruled out by imaging at screening;
10. Prior to starting the study treatment, there are:

    1. Poorly controlled diabetes (fasting blood glucose ≥ 13.3 mmol/L)
    2. Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
    3. History of hypertensive crisis or hypertensive encephalopathy
11. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening; Infusion-related thrombosis was excluded.
12. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). Patients who had received treatment for brain metastases (radiotherapy or surgery; Patients who had stopped radiotherapy and surgery 2 weeks before the first dose), and the long diameter of brain metastases < 10mm and stable brain metastases were eligible for inclusion. Patients with cancerous meningitis (meningeal metastasis) were excluded even if they were treated and judged to be stable.
13. Patients with pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage;
14. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any excipients of BL-B01D1;
15. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 103 IU/ml) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > detection limit);
17. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
18. Participated in another clinical trial within 4 weeks before the first dose (calculated from the time of the last dose);
19. Persons who have a history of psychotropic drug abuse and cannot be abstinent or have mental disorders;
20. Any other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B003.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, MB, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China